CLINICAL TRIAL: NCT04167072
Title: Scheduled Stent Removal vs Observation in Patients Undergoing EUS-guided Gallbladder Drainage. A Randomized Clinical Trial.
Brief Title: Observation vs Early Removal of LAMS in EUS Guided Cholecystoenterostomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected difficulties recruiting and following patients
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Antonio Mendoza-Ladd, Assistant Professor of Medicine/Director of Endoscopy, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20025
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Cholecystitis, Acute; Cholecystitis; Gallstone
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scheduled removal (Experimental): This group involves patients who will have the LAMS removed immediately after all the stones have been cleared from the gallbladder
  Interventions: Procedure: Stent removal
- Observation (Active Comparator): This group involves patients who will be followed closely for 1 year after all the stones have been removed from the gallbladder. These patients will keep the stent in place for 1 year and at that time the patients will be offered removal of the stent.
  Interventions: Procedure: Stent removal

INTERVENTIONS:
Procedure: Stent removal — This is a procedural intervention in which the stent will be removed via endoscopy.

SUMMARY:
The study will compare the outcomes of patients with gallstone related cholecystitis who are poor surgical candidates undergoing EUS guided cholecystoenterostomy via a lumen apposing metal stent (LAMS).

DETAILED DESCRIPTION:
The study will include patients with stone related cholecystitis that are not adequate surgical candidates that will be treated with EUS guided cholecystoenterostomy with endoscopic stone extraction. Patients will be randomized to stent removal immediately after gallstones have been removed or to observation for 1 year with the stent in place. Outcomes to be measured include recurrence of stone disease and rate of complications from the procedure in both groups

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-100 years or age
2. Both genders
3. Diagnosis of acute cholecystitis by TG13 criteria.
4. Patients who are able to give consent
5. Patients who are deemed poor surgical candidates for cholecystectomy by the surgical/medical team.

Exclusion Criteria:

1. Unable to provide informed consent
2. Cardiorespiratory dysfunction that precludes sedation
3. Pregnant females
4. Presence of ascites (distance between duodenum and GB > 1 cm) and/or coagulopathy (INR > 3, PLT <20K)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of GB findings | 1 year
  To compare the recurrence of GB findings in patients undergoing EUS guided GB drainage with a lumen-apposing metal stent(LAMS) assigned to scheduled stent removal vs those assigned to long-term observation only.

SECONDARY OUTCOMES:
Rate of adverse events related to LAMS | 1 year
  To compare the rate of LAMS related adverse events in these two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No